CLINICAL TRIAL: NCT02465853
Title: Clinical Outcome in Subacute Stroke Patients With Hemiplegic Shoulder Pain and Rotator Cuff Injuries After Hyaluronic Acid Injection
Brief Title: Hemiplegic Shoulder Pain and Rotator Cuff Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMRPG8C0771
Record Dates: First submitted 2014-12-16; First posted 2015-06-09 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2016-08

CONDITIONS: Shoulder Pain; Stroke; Rotator Cuff Injuries
Keywords: hemiplegic shoulder pain; quality of Life; stroke
MeSH Terms: conditions — Shoulder Pain; Stroke; Rotator Cuff Injuries | interventions — Hyaluronic Acid; Sodium Chloride; Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (Placebo Comparator): Injection 0.9% Physiological saline solution<2.5 ml and physical therapy and occupational therapy
  Interventions: Drug: Physiological saline solution; Other: physical therapy and occupational therapy
- Hyaluronic Acid (Experimental): injection Hyaluronic Acid 2.5ml and physical therapy and occupational therapy
  Interventions: Drug: Hyaluronic Acid; Other: physical therapy and occupational therapy

INTERVENTIONS:
Drug: Hyaluronic Acid — Injection Hyaluronic Acid in the experimental group
  Other Names: sodium hyaluronate
  Arms: Hyaluronic Acid
Drug: Physiological saline solution — Injection 0.9% Physiological saline solution<1.0 ml
  Other Names: saline
  Arms: Placebo group
Other: physical therapy and occupational therapy — rehabilitation

SUMMARY:
Hemiplegic shoulder pain (HSP) is one of most complications after stroke. HSP would impede rehabilitation programs and the motor recovery of affected upper extremity. HSP was associated with impaired daily life activities and prolong hospital stay after stroke. Therefore, effective managements is important in stroke patients with HSP. Rotator cuffs injuries are related to HSP. Clinically, hyaluronic acid (HA) is used for rotator cuff injuries. Previous researchers reported that HA could provide pain relief, improved motion, and increased daily activities. In this study, fifty subacute stoke patients will be enrolled. These patients will be allocated into group A and B randomly. The patients in group A received HA injection while patients in group B received normal saline injection. Patients from both groups received injection for 3 times each on the 1st, 2nd, 3rd week. All the patients will still receive rehabilitation programs of physical therapy and occupational therapy. Each patient will receive physical, sonographic examinations, and stroke Specific Quality of Life Scale (SSQOL). The aims of this study are to investigate the benefits of HA injection on pain relief, motor function recovery, and life quality in subacute stroke patients with HSP before and after HA injection.

DETAILED DESCRIPTION:
In this study, a two-year program is expected to receive a total cases of 50 subacute stroke patients with hemiplegic shoulder pain. The patients are randomly divided into two groups. In experimental group, the patients (25 people) will accept the shoulder hyaluronic acid injections for pain management. In control group, the patients (25 people) will receive 0.9% physiological saline injections. All participants will receive total 3 times shoulder injections at the 1st, 2nd, 3rd week. Except shoulder injections, stroke patients may receive regular rehabilitation program including physical therapy and occupational therapy. All measurements including shoulder sonography, physical examinations, and the questionnaire for life quality (SSQOL) will be conducted before the first injection, after completing shoulder injection, and 3/6 months after shoulder injection. Shoulder sonography is used to investigate shoulder soft tissue condition of hemiplegic shoulder including biceps tendon, infraspinatus tendon, supraspinatus tendon, subscapularis tendon, and subdeltoid bursa in this study. The physical examination includes all shoulder motion plane, shoulder sensory (light touch, pinprick, and position sense) and motor function (Fual Meyer scale and brunnstrom motor recovery stage), shoulder spasticity measured by modified Ashworth scale, and hemiplegic shoulder pain by visual analog scale. The investigators use Stroke Specific Quality of Life Scale to evaluate the quality of life in stroke patients with HSP. In this study, the investigators want to explore the short and long term effects of HA injection on pain relief, motor function recovery, and life quality in stroke patients with HSP.

ELIGIBILITY:
Inclusion Criteria:

* The subacute stroke patients with hemiplegic shoulder pain

Exclusion Criteria:

* previous shoulder pain or injury in recent 6 months
* local infection near the injection area
* shoulder arthropathy
* systemic neuromuscular disease;
* severe cardiovascular or pulmoanry disease
* impaired cognition function leading to poor communication

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-01; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
the change from baseline on hemiplegic shoulder sonography | 1 week , 4th week, 3 month and 6 month
  use sonographic to investigate the soft tissues surrounding the hemiplegic shoulder

SECONDARY OUTCOMES:
shoulder range of motion | 1 week , 4th week, 3 month and 6 month
  goniometer Shoulder abduction 0-180, flex 0-180, ext 0-60, internal rotation 0-90, external rotation 0-90
Quality of Life | 1 week , 4th week, 3 month and 6 month
  Stroke Specific Quality of Life Scale questionnaire
shoulder sensory | 1 week , 4th week, 3 month and 6 month
  light touch, pin prick, position sense
shoulder pain | 1 week , 4th week, 3 month and 6 month
  visual analog scale
shoulder spasticity | 1 week , 4th week, 3 month and 6 month
  modified Ashworth scale
motor function | 1 week , 4th week, 3 month and 6 month
  Fual Meyer scale, brunnstrom motor recovery stage

CONTACTS AND LOCATIONS:
Overall Officials: Huang Yu Chi, Bachelor, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- ChangGungMH, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
no available now

REFERENCES:
- [Background] Najenson T, Yacubovich E, Pikielni SS. Rotator cuff injury in shoulder joints of hemiplegic patients. Scand J Rehabil Med. 1971;3(3):131-7. No abstract available. PMID 5156175
- [Background] Griffin J, Reddin G. Shoulder pain in patients with hemiplegia. A literature review. Phys Ther. 1981 Jul;61(7):1041-5. doi: 10.1093/ptj/61.7.1041. No abstract available. PMID 6166017
- [Background] Bohannon RW, Larkin PA, Smith MB, Horton MG. Shoulder pain in hemiplegia: statistical relationship with five variables. Arch Phys Med Rehabil. 1986 Aug;67(8):514-6. PMID 3741075
- [Background] Turner-Stokes L, Jackson D. Shoulder pain after stroke: a review of the evidence base to inform the development of an integrated care pathway. Clin Rehabil. 2002 May;16(3):276-98. doi: 10.1191/0269215502cr491oa. PMID 12017515
- [Background] Snels IA, Dekker JH, van der Lee JH, Lankhorst GJ, Beckerman H, Bouter LM. Treating patients with hemiplegic shoulder pain. Am J Phys Med Rehabil. 2002 Feb;81(2):150-60. doi: 10.1097/00002060-200202000-00013. PMID 11807352
- [Background] Van Ouwenaller C, Laplace PM, Chantraine A. Painful shoulder in hemiplegia. Arch Phys Med Rehabil. 1986 Jan;67(1):23-6. PMID 3942479
- [Background] Gilmore PE, Spaulding SJ, Vandervoort AA. Hemiplegic shoulder pain: implications for occupational therapy treatment. Can J Occup Ther. 2004 Feb;71(1):36-46. doi: 10.1177/000841740407100108. PMID 15015899
- [Background] Snels IA, Beckerman H, Twisk JW, Dekker JH, Peter De Koning, Koppe PA, Lankhorst GJ, Bouter LM. Effect of triamcinolone acetonide injections on hemiplegic shoulder pain : A randomized clinical trial. Stroke. 2000 Oct;31(10):2396-401. doi: 10.1161/01.str.31.10.2396. PMID 11022070
- [Background] Parker VM, Wade DT, Langton Hewer R. Loss of arm function after stroke: measurement, frequency, and recovery. Int Rehabil Med. 1986;8(2):69-73. doi: 10.3109/03790798609166178. PMID 3804600
- [Background] Wanklyn P, Forster A, Young J. Hemiplegic shoulder pain (HSP): natural history and investigation of associated features. Disabil Rehabil. 1996 Oct;18(10):497-501. doi: 10.3109/09638289609166035. PMID 8902421
- [Background] Roy C SM, Hill L. Shoulder pain in acutely admitted hemiplegics. Clinical Rehabilitation. 1994;8:334-340
- [Background] Lo SF, Chen SY, Lin HC, Jim YF, Meng NH, Kao MJ. Arthrographic and clinical findings in patients with hemiplegic shoulder pain. Arch Phys Med Rehabil. 2003 Dec;84(12):1786-91. doi: 10.1016/s0003-9993(03)00408-8. PMID 14669184
- [Background] Ikai T, Tei K, Yoshida K, Miyano S, Yonemoto K. Evaluation and treatment of shoulder subluxation in hemiplegia: relationship between subluxation and pain. Am J Phys Med Rehabil. 1998 Sep-Oct;77(5):421-6. doi: 10.1097/00002060-199809000-00012. PMID 9798835
- [Background] Poulin de Courval L, Barsauskas A, Berenbaum B, Dehaut F, Dussault R, Fontaine FS, Labrecque R, Leclerc C, Giroux F. Painful shoulder in the hemiplegic and unilateral neglect. Arch Phys Med Rehabil. 1990 Aug;71(9):673-6. PMID 2375673
- [Background] Ada L, Goddard E, McCully J, Stavrinos T, Bampton J. Thirty minutes of positioning reduces the development of shoulder external rotation contracture after stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2005 Feb;86(2):230-4. doi: 10.1016/j.apmr.2004.02.031. PMID 15706548
- [Background] Griffin A, Bernhardt J. Strapping the hemiplegic shoulder prevents development of pain during rehabilitation: a randomized controlled trial. Clin Rehabil. 2006 Apr;20(4):287-95. doi: 10.1191/0269215505cr941oa. PMID 16719027
- [Background] Ada L, Foongchomcheay A, Canning C. Supportive devices for preventing and treating subluxation of the shoulder after stroke. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003863. doi: 10.1002/14651858.CD003863.pub2. PMID 15674917
- [Background] Chae J, Yu DT, Walker ME, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Frost FS, Grill JH, Fang ZP. Intramuscular electrical stimulation for hemiplegic shoulder pain: a 12-month follow-up of a multiple-center, randomized clinical trial. Am J Phys Med Rehabil. 2005 Nov;84(11):832-42. doi: 10.1097/01.phm.0000184154.01880.72. PMID 16244520
- [Background] Chantraine A, Baribeault A, Uebelhart D, Gremion G. Shoulder pain and dysfunction in hemiplegia: effects of functional electrical stimulation. Arch Phys Med Rehabil. 1999 Mar;80(3):328-31. doi: 10.1016/s0003-9993(99)90146-6. PMID 10084443
- [Background] Shibata Y, Midorikawa K, Emoto G, Naito M. Clinical evaluation of sodium hyaluronate for the treatment of patients with rotator cuff tear. J Shoulder Elbow Surg. 2001 May-Jun;10(3):209-16. doi: 10.1067/mse.2001.113501. PMID 11408900
- [Background] Blair B, Rokito AS, Cuomo F, Jarolem K, Zuckerman JD. Efficacy of injections of corticosteroids for subacromial impingement syndrome. J Bone Joint Surg Am. 1996 Nov;78(11):1685-9. doi: 10.2106/00004623-199611000-00007. PMID 8934482
- [Background] Vecchio PC, Hazleman BL, King RH. A double-blind trial comparing subacromial methylprednisolone and lignocaine in acute rotator cuff tendinitis. Br J Rheumatol. 1993 Aug;32(8):743-5. doi: 10.1093/rheumatology/32.8.743. PMID 8348279
- [Background] Plafki C, Steffen R, Willburger RE, Wittenberg RH. Local anaesthetic injection with and without corticosteroids for subacromial impingement syndrome. Int Orthop. 2000;24(1):40-2. doi: 10.1007/s002640050010. PMID 10774861
- [Background] Akgun K, Birtane M, Akarirmak U. Is local subacromial corticosteroid injection beneficial in subacromial impingement syndrome? Clin Rheumatol. 2004 Dec;23(6):496-500. doi: 10.1007/s10067-004-0930-7. PMID 15278758
- [Background] Penning LI, de Bie RA, Walenkamp GH. The effectiveness of injections of hyaluronic acid or corticosteroid in patients with subacromial impingement: a three-arm randomised controlled trial. J Bone Joint Surg Br. 2012 Sep;94(9):1246-52. doi: 10.1302/0301-620X.94B9.28750. PMID 22933498
- [Background] Iwata H. Pharmacologic and clinical aspects of intraarticular injection of hyaluronate. Clin Orthop Relat Res. 1993 Apr;(289):285-91. PMID 8472428
- [Background] Meloni F, Milia F, Cavazzuti M, Doria C, Lisai P, Profili S, Meloni GB. Clinical evaluation of sodium hyaluronate in the treatment of patients with sopraspinatus tendinosis under echographic guide: experimental study of periarticular injections. Eur J Radiol. 2008 Oct;68(1):170-3. doi: 10.1016/j.ejrad.2007.11.001. Epub 2007 Dec 21. PMID 18096343
- [Background] Chou WY, Ko JY, Wang FS, Huang CC, Wong T, Wang CJ, Chang HE. Effect of sodium hyaluronate treatment on rotator cuff lesions without complete tears: a randomized, double-blind, placebo-controlled study. J Shoulder Elbow Surg. 2010 Jun;19(4):557-63. doi: 10.1016/j.jse.2009.08.006. Epub 2009 Dec 5. PMID 19963403
- [Background] Byun SD, Park DH, Choi WD, Lee ZI. Subacromial Bursa Injection of Hyaluronate with Steroid in Patients with Peri-articular Shoulder Disorders. Ann Rehabil Med. 2011 Oct;35(5):664-72. doi: 10.5535/arm.2011.35.5.664. Epub 2011 Oct 31. PMID 22506189
- [Background] Blaine T, Moskowitz R, Udell J, Skyhar M, Levin R, Friedlander J, Daley M, Altman R. Treatment of persistent shoulder pain with sodium hyaluronate: a randomized, controlled trial. A multicenter study. J Bone Joint Surg Am. 2008 May;90(5):970-9. doi: 10.2106/JBJS.F.01116. PMID 18451387
- [Background] Itokazu M, Matsunaga T. Clinical evaluation of high-molecular-weight sodium hyaluronate for the treatment of patients with periarthritis of the shoulder. Clin Ther. 1995 Sep-Oct;17(5):946-55. doi: 10.1016/0149-2918(95)80072-7. PMID 8595646
- [Background] Ko JY, Wang FS, Huang HY, Wang CJ, Tseng SL, Hsu C. Increased IL-1beta expression and myofibroblast recruitment in subacromial bursa is associated with rotator cuff lesions with shoulder stiffness. J Orthop Res. 2008 Aug;26(8):1090-7. doi: 10.1002/jor.20631. PMID 18327798